CLINICAL TRIAL: NCT01470547
Title: Portal Vein Thrombosis Relevance On Liver Cirrhosis: Italian Venous Thrombotic Events Registry
Acronym: PRO-LIVER
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Collaborators: University of Pavia (Other)
Responsible Party: Principal Investigator, Francesco Violi, Prof., University of Roma La Sapienza
Other Study IDs: SIMI PRO-LIVER
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Liver Cirrhosis; Portal Vein Thrombosis
Keywords: Liver Cirrhosis; Portal Vein Thrombosis; Cirrhosis Complications; Registry; Italian
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum samples (in ancillary study)
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The portal vein thrombosis (PVT) can complicate medical conditions like liver cirrhosis (LC), neoplasms, myeloproliferative diseases, thrombophilic genotypes, infections, inflammatory diseases, trauma and surgery. LC is an important predisposing disease and is responsible for about 20% of all cases. However, data regarding the PVT in cirrhosis are insufficient.

Early studies have shown that, in absence of hepatocellular carcinoma (HCC), the PVT can occur in approximately 10% of cirrhotic patients.

Most of studies are in support of a prevalence between 5 and 20% of patients with LC. A study in transplant recipients, has documented that in variable etiology cirrhosis, the PVT was present in 15.7% of patients, a higher percentage was found in patients with liver cancer (34.8%), while primary biliary cirrhosis (7.9%) and sclerosing cholangitis (3.6%) are less frequently complicated by PVT.

The PVT development is due to stagnation in the portal circulation, but alterations in the sense of inherited or acquired pro-coagulant may favor its appearance.

The causal association of PVT with bleeding and bowel infarction suggests that the PVT may reduce survival in cirrhosis, but data are lacking on this issue. It is also not known whether asymptomatic patients with PVT have a different survival compared to cirrhotic patients without PVT. Further studies should be conducted to clarify this issue.

Likewise, prospective studies are needed to better identify risk factors predisposing to PVT in LC patients as well as to clarify the relationship between cirrhosis severity and PVT. The impact of PVT on the natural history of cirrhosis is an issue today still debated.

The PVT not only favour life-threatening complications (gastrointestinal bleeding and mesenteric thrombosis) but could also contribute to a deterioration of liver function by reducing portal flow. Obtaining such information would be of crucial importance considering that the evidence of increased mortality related to PVT in liver cirrhosis may indicate the need for randomized controlled trials to clarify the potential effectiveness of anticoagulant therapy to improve the survival.

To this purpose it's proposed to establish an Italian register of patients with cirrhosis. In the second phase of the project is planned a 2-years follow-up program in order to assess whether the PVT be an additional risk factor for mortality or deterioration of the natural history in patients with cirrhosis.

DETAILED DESCRIPTION:
Study Design: Prospective Longitudinal Study.

The investigators planned to assess at baseline and at scheduled follow up visits:

* Medical history collection with thrombosis risk factors evaluation;
* Clinical parameters collection;
* Upper abdomen ultrasound and portal district echo color doppler to evaluate the presence of PVT;
* Esophagogastroduodenoscopy;
* Routine blood samples collection with plasma and urine storage;

At every follow up visit will be evaluated all relevant clinical events and will be recorded all treatments received during the follow-up period.

Sample Size: The investigators plan to include in the study n = 1100 patients. The sample size was calculated assuming an expected prevalence of 18% at time zero, and in order to obtain a confidence interval 95% to prevail at time zero whose distance from the edge is less than or equal to 3%.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis of any etiology and severity (including HCC)
* Signed Written Informed Consent

Exclusion Criteria:

* Extrahepatic neoplasms

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Liver cirrhosis patients
Sampling Method: Probability Sample
Enrollment: 753 (Actual)
Dates: Start 2012-04; Primary Completion 2017-04 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
PVT prevalence | 1 year
  To estimate the prevalence of PVT evaluated by US with power-doppler in a cohort of patients with liver cirrhosis of any etiology and severity.

SECONDARY OUTCOMES:
Thrombotic Events | 2 years
  Occurrence of thrombotic complications (deep vein and portal vein thrombosis)
Mortality | 2 Years
  Overall mortality in a cohort of cirrhotic patients
Cirrhosis Complications | 2 Years
  Occurence of other cirrhosis-related complications (previous refractory ascites or hepatic encephalopathy; onset or progression of oesophageal varices, ascites or refractory ascites, jaundice, onset of liver cancer, infections, spontaneous bacterial peritonitis, onset of hepato-renal or hepato-pulmonary syndrome)
Bleeding | 2-4 years
  Occurrence of digestive or other mjor or minor bleeding events in relation to platelet count and/or PT-INR

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Violi, MD, Study Chair — Divisione di Prima Clinica Medica - Sapienza University of Rome and SIMI; Gino R Corrazza, MD, Study Chair — Fondazione IRCCS Policlinico San Matteo and SIMI
Locations (2):
- Italy (2):
  - Sapienza - University of Rome, Rome, RM
  - Società Italiana di Medicina Interna, Rome, RM

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] D'Amico T, Miglionico M, Cangemi R, Romiti GF, De Fabrizio B, Fasano S, Recchia F, Stefanini L, Raparelli V, Violi F, Basili S; P. R. O.-LIVER Collaborators. Neutrophil-lymphocyte ratio is associated with worse outcomes in patients with cirrhosis: insights from the PRO-LIVER Registry. Intern Emerg Med. 2025 Aug;20(5):1371-1380. doi: 10.1007/s11739-025-03955-x. Epub 2025 May 20. PMID 40392481
- [Derived] Violi F, Corazza GR, Caldwell SH, Perticone F, Gatta A, Angelico M, Farcomeni A, Masotti M, Napoleone L, Vestri A, Raparelli V, Basili S; PRO-LIVER Collaborators. Portal vein thrombosis relevance on liver cirrhosis: Italian Venous Thrombotic Events Registry. Intern Emerg Med. 2016 Dec;11(8):1059-1066. doi: 10.1007/s11739-016-1416-8. Epub 2016 Mar 30. PMID 27026379
- See also: Società Italiana di Medicina Interna — http://www.simi.it
- See also: Preliminary data — https://www.ncbi.nlm.nih.gov/pubmed/27026379